CLINICAL TRIAL: NCT05167929
Title: Effects of a Culturally-tailored Personal Self-Determination Enhancement Intervention for People With Mild Intellectual Disabilities and Their Caregivers in Hong Kong - A Randomised Controlled Trial
Brief Title: Self-determination Enhancement Group for Adults With Mild Intellectual Disability and Their Caregivers in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong King Shui, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24617019
Record Dates: First submitted 2021-11-22; First posted 2021-12-22 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Intellectual Disability, Mild
Keywords: Self-determination enhancement;; intellectual disability;; culturally-tailored group;; Chinese societies;; randomised controlled trial
MeSH Terms: conditions — Intellectual Disability; Lymphoma, Follicular | interventions — Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental)
  Interventions: Behavioral: Self-determination Enhancement Group
- Intervention PLUS Group (Experimental)
  Interventions: Behavioral: Self-determination Enhancement Plus Group
- Comparison Group (Active Comparator)
  Interventions: Behavioral: Leisure activity group

INTERVENTIONS:
Behavioral: Self-determination Enhancement Group — The self-determination enhancement group - Each group has eight participants. There will be 10 sessions per group and each session will last 1.5 hours.
  Arms: Intervention Group
Behavioral: Self-determination Enhancement Plus Group — The self-determination enhancement PLUS group - Each group has eight participants and their caregivers. There will be 10 sessions per group and each session will last 1.5 hours. Meanwhile, their caregivers will attend four sessions separately and each session will last 1.5 hours.
  Arms: Intervention PLUS Group
Behavioral: Leisure activity group — Leisure activity group - Leisure activity group is the comparison group. Each group will consist of eight adults with mild intellectual disability. There will be 10 sessions for the group and each session will last for 1.5 hours.
  Arms: Comparison Group

SUMMARY:
Background Self-determination is regarded as an adult outcome for people with intellectual disability (ID). Students with ID in western countries learn self-determination knowledge and skills through the systematic curriculum in schools. However, the curriculum for adults with ID is still underdeveloped in the West. In Hong Kong, the self-determination curriculum is rarely available in any setting.

Objective The proposed study aims to develop a culturally-tailored self-determination enhancement group intervention for adults with ID and to evaluate its effectiveness.

Method The proposed study will consist of two phases. Phase one will develop the protocol for the self-determination enhancement intervention and establish its implementation fidelity through a panel review and pilot study. This phase will last eight months. Phase two will adopt a randomised controlled trial with pre-test, post-test and three-month follow-up. A total of 120 participants will be randomly assigned to three conditions: Self-determination enhancement group, Self-determination enhancement PLUS group (+ parents' involvement) and leisure activity group as a control condition. Five groups will be organised for each of the three conditions over 18 months. There will be 10 sessions per group covering the self-determination core components such as self-understanding, goal-setting and attaining, self-regulating and plan adjusting. Components for parents include understanding self-determination and skills in supporting people with ID to exercise self-determination through positive interaction. Validated instruments in Chinese will be filled in by participants. Statistical analyses will be conducted to examine if the effectiveness of this group intervention can be found and sustained over a three-month period, and the magnitude of change in self-determination competencies and quality of life.

Implications The proposed study is the first evidence-based local study aimed at examining a culturally-tailored self-determination enhancement intervention for people with ID. If the intervention demonstrated as effective, it will be used or modified for use with Chinese-speaking people with ID in different parts of the world.

ELIGIBILITY:
Inclusion Criteria:

* Chinese people who have mild intellectual disability (i.e., assessed in their most recent psychological report)
* Aged 18 or above
* Able to master basic comprehension and verbal communication skills
* Willing to complete the group intervention.

Exclusion Criteria:

* Those who demonstrate severe challenging behaviours will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Changes of self-determination competence level | Pretest (T0) - baseline; posttest (T1) - after the completion of the intervention (3 months later from the pretest); and follow-up test (T2) (3 months later from the posttest)
  The AIR Self-Determination Scale: the Chinese Version (AIR SDS-C) (Wong, Wong, Zhuang & Liu, 2017) will be used. This is a 24-items, 5-point Likert-scale questionnaire to measure the self-determination of people with intellectual disability

SECONDARY OUTCOMES:
Changes of personal well-being questionnaire | Pretest (T0) - baseline; posttest (T1) - after the completion of the intervention (3 months later from the pretest); and follow-up test (T2) (3 months later from the posttest)
  The Personal Well-being: Intellectual Disability (Cantonese) 3rd Edition (PWI-C). This is an 8-item, 5-point Likert-scale questionnaire used to measure the subjective well-being of people with intellectual disability

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis KS WONG, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong PKS. Study Protocol for a Randomized Controlled Trial Evaluating the Effectiveness of a Group-Based Self-Determination Enhancement Intervention for Adults with Mild Intellectual Disability and Their Caregivers. Int J Environ Res Public Health. 2022 Feb 4;19(3):1763. doi: 10.3390/ijerph19031763. PMID 35162786